CLINICAL TRIAL: NCT06073964
Title: Gender Based Violence and the Level of Utilization of the 'Trauma Resilience & Understanding Self-help Therapy' Among Formerly Internally Displaced Persons Living in Lira District, Northern Uganda
Brief Title: GBV, Primary Trauma & Trauma Resilience & Understanding Self-help Therapy Utilization in Uganda
Acronym: GBV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kampala International University (Other)
Collaborators: Dutch Research Council (WOTRO Impact and Innovation Grants-2020), The Netherlands (Unknown); Leiden University (Other); Globalization Accessibility Innovation and Care Research Collaborative Network (Unknown)
Responsible Party: Principal Investigator, Jimmy Ben Forry, Principal Investigator, Kampala International University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KIU-2022-173
Record Dates: First submitted 2023-09-26; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Domestic Violence; Psychological Distress; Post-Traumatic Stress Disorder; Suicidality
Keywords: formerly Internally Displaced Persons; Gender Based Violence; Trauma Resilience & Understanding Self-help Therapy; Uganda
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRUST Intervention group (Experimental): Formerly Internally Displaced Persons living in Lira district, northern Uganda afflicted with primary trauma and experiencing domestic violence will be trained in the community-based utilization of the 'Trauma Resilience & Understanding Self-help Therapy'.
  Interventions: Behavioral: Trauma Resilience & Understanding Self-help Therapy
- Control group (No Intervention): Age and gender cross-matched formerly Internally Displaced Persons living in Lira district, northern Uganda afflicted with primary trauma and experiencing domestic violence will not be trained in the community-based utilization of the 'Trauma Resilience & Understanding Self-help Therapy'.

INTERVENTIONS:
Behavioral: Trauma Resilience & Understanding Self-help Therapy — A self-help psychosocial therapeutic intervention requiring one to undergo a basic training in its community-based utilization.
  Arms: TRUST Intervention group

SUMMARY:
The goal of this community-based interventional study was to determine the effectiveness of the 'Trauma Resilience & Understanding Self-help Therapy' (TRUST) in managing domestic violence & primary trauma among formerly Internally Displaced Persons (fIDPs) in northern Uganda. The main questions it aimed to answer were:

* What was the level of utilization and short-term effects of the TRUST intervention on the experiences of domestic violence and high levels of primary trauma among fIDPs living in northern Uganda who would have been using TRUST within their communities after completing the training in the community-based TRUST utilization?
* What were the clinical indications of the TRUST intervention and psychological operators among fIDPs living in northern Uganda who would have been using TRUST within their communities to manage their experiences of domestic violence and high levels of primary trauma? Participants found to have experienced domestic violence in the last one year and were having high levels of primary trauma were randomly assigned to the intervention group that was trained in the utilization of the TRUST within their communities and then followed up for 12 weeks (TRUST group).

The investigators then compared the results obtained from the TRUST group with those attained from an age and gender cross-matched control group of fIDPs who were not trained in the utilization of the TRUST within their communities (Control group). This was done to see if the community-based utilization of the TRUST intervention changed the levels of primary trauma & experiences of domestic violence among its users (TRUST group) when compared to the non-users (Control group).

DETAILED DESCRIPTION:
An indigenous rebel outfit waged a decades' civil war in eastern and northern Uganda until the early 2000s. This rebellion resulted in forceful internal displacement of most of the local population leading to unwarranted misery. In the aftermath of this rebellion, the internally displaced returned to their areas of origin. However, a significant proportion of these formerly internally displaced persons (fIDPs) have since then been plagued with a plethora of adversities including high levels of primary trauma, frequent experiences of domestic violence and impaired social economic resilience (SER) levels. A newly developed psychosocial therapeutic intervention called the 'trauma resilience & understanding self-help therapy' (TRUST) was revealed to be qualitatively effective in managing high levels of primary trauma, experiences of domestic violence and poor SER levels among refugees and fIDPs. However, the quantitative effectiveness of TRUST and the psychological operators among the fIDPs and refugees within which it is grounded still remain a scientific mystery. Hence, an appropriate prospective community-based cohort research study was conducted to this effect. The investigators carried out a descriptive community-based prospective study from November 2022 to March 2023 among 284 randomly recruited adults who were fIDPs living in northern Uganda using quantitative data collection techniques in natural experiments conducted via repeated assessments. The resultant data were analyzed using univariate, bivariate and multivariate linear, logistic and Poisson regression as well as determining the effect sizes of the community-based utilization of TRUST on the high levels of primary trauma, experiences of domestic violence and poor SER levels among fIDPs living in northern Uganda. These findings were compared with those obtained among a randomly selected control group of fIDPs living in northern Uganda who were cross-matched according to their age and gender, were experiencing high levels of primary trauma and domestic violence as well as poor SER levels and had not been trained in the community-based utilization of TRUST.

ELIGIBILITY:
Inclusion Criteria:

* All formerly Internally Displaced Persons who will be 18 years or older and who will be residing in the sub-counties of Agweng, Barr and Ogur in Lira district, northern Uganda at the time of data collection.
* All formerly Internally Displaced Persons who will be residing in Agweng and Ogur sub-counties at the time of data collection and who previously participated in the study that culminated in the development of the TRUST intervention in Lira district, northern Uganda.
* All formerly Internally Displaced Persons who will be residing in Agweng, Barr and Ogur sub-counties in Lira district, northern Uganda at the time of data collection and who will screen positive for domestic violence, psychological distress and PTSD.

Exclusion Criteria:

* All formerly Internally Displaced Persons who will be residing in the sub-counties of Agweng, Barr and Ogur in Lira district, northern Uganda and who will have clinically significant or overt baseline signs and symptoms of physical illnesses or other psychiatric disorders which are unrelated to primary trauma or domestic violence.
* All formerly Internally Displaced Persons who will be residing in the sub-counties of Agweng, Barr and Ogur in Lira district, northern Uganda at the time of data collection and who will have significantly severe hearing and speech impediments.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Rate of Domestic Violence Experiences | Pilot Study, Baseline/Pre-TRUST Training (After 1 month from the pilot study), Post-TRUST Training (After 6 weeks) & Post-TRUST Utilization (After 12 weeks)
  Change in frequency of experiences assessed using the Assessment Screen to Identify Survivors' Toolkit for Gender Based Violence Scale.
Prevalence of Psychological Distress | Pilot Study, Baseline/Pre-TRUST Training (After 1 month from the pilot study), Post-TRUST Training (After 6 weeks) & Post-TRUST Utilization (After 12 weeks)
  Change in severity of symptoms assessed using the Refugee Health Sceener-15 Scale.
Prevalence of Post-Traumatic Stress Disorder | Pilot Study, Baseline/Pre-TRUST Training (After 1 month from the pilot study), Post-TRUST Training (After 6 weeks) & Post-TRUST Utilization (After 12 weeks)
  Change in severity of symptoms assessed using the Impact of Events Scale-Shorter Revised Scale & the Mini International Neuropsychiatric Interview guide module H for Post-Traumatic Stress Disorder.
Prevalence of Suicidality Risk | Pilot Study, Baseline/Pre-TRUST Training (After 1 month from the pilot study), Post-TRUST Training (After 6 weeks) & Post-TRUST Utilization (After 12 weeks)
  Change in levels of risk assessed using the Mini International Neuropsychiatric Interview guide module B for Suicidality Risk.

SECONDARY OUTCOMES:
Prevalence of Poor Social Economic Resilience Levels | Pilot Study, Baseline/Pre-TRUST Training (After 1 month from the pilot study), Post-TRUST Training (After 6 weeks) & Post-TRUST Utilization (After 12 weeks)
  Change in levels of impairment assessed using the Social Economic Resilience Scale-Shorter version.

OTHER OUTCOMES:
Percentage of Participants with impaired Psychological Indicators | Pilot Study, Baseline/Pre-TRUST Training (After 1 month from the pilot study), Post-TRUST Training (After 6 weeks) & Post-TRUST Utilization (After 12 weeks)
  Changes in mental state examination findings assessed via a comprehensive clinical neuropyschiatric evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy B Forry, MMed Psych, Principal Investigator — Kampala International University
Locations (1):
- Kampala International University, Bushenyi, Southwestern, Uganda

IPD SHARING:
Plan to Share IPD: No
This is due to the sensitive nature of the data and their legal implications.

REFERENCES:
- [Result] Forry, J. B., Kirabira, J., Akimana, B., Nakawuki, M., Gumisiriza, N., Ssebuufu, R., & Ashaba, S. (2022). Gender-based violence and its determinants during the COVID-19 lockdown in a low-income country: a cross-sectional survey. Journal of gender-based violence, 1-19.
- See also: Background Peer-reviewed Published Article — https://bristoluniversitypressdigital.com/view/journals/jgbv/aop/article-10.1332-239868021X16460622083652/article-10.1332-239868021X16460622083652.xml